CLINICAL TRIAL: NCT00103051
Title: Phase II Study With Gefitinib (Sequentially) Following Gemcitabine/Cisplatin as Induction Regimen for Patients With Stage IIIA N2 NSCLC
Brief Title: Gemcitabine, Cisplatin, and Gefitinib in Treating Patients Who Are Undergoing Surgery for Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-08013; EORTC-08013; 2004-001332-23 (EudraCT Number)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gefitinib; Gemcitabine; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: gefitinib
Drug: gemcitabine hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine and cisplatin together with gefitinib before surgery may shrink the tumor so it can be removed.

PURPOSE: This phase II trial is studying how well giving gemcitabine and cisplatin together with gefitinib works in treating patients who are undergoing surgery for stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the therapeutic activity of neoadjuvant induction therapy comprising gemcitabine, cisplatin, and gefitinib in patients with stage IIIA non-small cell lung cancer undergoing surgery.

Secondary

* Determine the safety profile of this regimen in these patients.
* Determine the stage downsizing and complete resectability rate in patients with no progressive disease who undergo surgery after treatment with this regimen.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive induction therapy comprising gemcitabine IV over 30 minutes on days 1, 8, 22, 29, 43, and 50; cisplatin IV over 3-6 hours on days 2, 23, and 44; and oral gefitinib once daily on days 51-79. Treatment continues in the absence of disease progression or unacceptable toxicity. Within 2-7 days after completion of induction therapy, patients with no progressive disease undergo tumor resection.

After completion of study treatment, patients are followed at least every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary non-small cell lung cancer (NSCLC)

  * Clinical stage IIIA by chest CT scan
  * Unresectable N2 disease by mediastinoscopy, mediastinotomy, thoracotomy, or video-assisted thoracic surgery
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Planning to undergo lobectomy or pneumonectomy after induction therapy
* No N3 or metastatic disease by physical exam, thoracic CT scan, bone scan, and CT scan or ultrasound of the liver and adrenal glands
* No pleural or pericardial effusion
* No superior vena cava syndrome
* No diffuse interstitial pulmonary fibrosis
* No signs or symptoms of CNS involvement

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.25 times ULN
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No medically uncontrolled congestive heart failure or angina pectoris
* No uncontrolled hypertension or arrhythmia
* No myocardial infarction within the past year

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Physically and mentally fit to receive gemcitabine- and cisplatin-containing chemotherapy
* Physiologically fit to undergo surgery
* No uncontrolled, active infection requiring IV antibiotics
* No history of hypersensitivity to gefitinib or any of its excipients
* No motor or sensory neurotoxicity ≥ grade 2
* No other primary malignancy within the past 5 years except carcinoma in situ of the cervix or adequately treated basal cell skin cancer

  * No prior melanoma, breast cancer, or renal cell cancer
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy for NSCLC
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent antiestrogen therapy
* Concurrent replacement steroids and antiemetic steroids allowed

Radiotherapy

* No prior radiotherapy for NSCLC

Surgery

* See Disease Characteristics
* No prior surgery for NSCLC

Other

* More than 1 month since prior and no concurrent investigational agents
* No other prior therapy for NSCLC
* No concurrent CYP3A4 inducers, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Barbiturates (e.g., phenobarbital)
  * Hypericum perforatum (St. John's wort)
* No concurrent systemic retinoids
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Complete response rate as measured by RECIST criteria prior to surgery

SECONDARY OUTCOMES:
Overall response rate as measured by RECIST criteria prior to surgery
Toxicity as assessed by CTC

CONTACTS AND LOCATIONS:
Overall Officials: Nico Van Zandwijk, MD, PhD, Study Chair — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands